CLINICAL TRIAL: NCT05152407
Title: MRB 0.3% Serum Effectiveness on 2 Early Clinical Markers of Photoinduced Cutaneous Aging: Actinic Lentigo and Actinic Keratosis A Single-center Clinical Study in Two Phases: First Phase: Randomized Double-blind Clinical Interventional Study Versus Placebo in Split Face or Split Skull Second Phase: Open-label Observational Clinical Study on the Entire Face or Skull
Brief Title: MRB 0.3% Serum Effectiveness on 2 Early Clinical Markers of Photoinduced Cutaneous Aging: Actinic Lentigo and Actinic Keratosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NAOS Institute of Life Science (Industry)
Responsible Party: Principal Investigator, JULIE TISSERAND, PhD, Project manager, NAOS Institute of Life Science
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3020_ILS-MIRORU20; ID RCB 2020-A02883-36 (Other: ANSM)
Record Dates: First submitted 2021-11-24; First posted 2021-12-09 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Actinic Keratosis; Actinic Lentigo
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active serum on right (Experimental): Right hemi face or skull will receive active serum (containing 0.3% MRB) / Left hemi face or skull will receive placebo serum for 6 months
  Interventions: Other: Topical application of MRB 0.3% serum and placebo serum (hemi face or skull)
- Active serum on left (Experimental): Left hemi face or skull will receive active serum (containing 0.3% MRB) / Right hemi face or skull will receive placebo serum for 6 months
  Interventions: Other: Topical application of MRB 0.3% serum and placebo serum (hemi face or skull)

INTERVENTIONS:
Other: Topical application of MRB 0.3% serum and placebo serum (hemi face or skull) — Serums will be topically applied twice a day (mornings and evenings).

SUMMARY:
The aim of this study is to evaluate effectiveness of a serum containing 0.3% of MRB, a cosmetic active ingredient, against actinic lentigo and actinic keratosis.

DETAILED DESCRIPTION:
Skin aging is an extremely complex multifactorial process that disrupts the functions and structure of epidermal and dermal cells and extracellular matrix components and has multiple causes including extrinsic phenomena (UV radiation, exposure to pollution, etc.).

It has important effects on the skin and is particularly apparent on the face. Indeed, sunlight, in particular ultraviolet light, is an important factor that contributes to cutaneous photoaging by inducing the photo-chronic generation of reactive oxygen species (ROS). Although skin has its own antioxidant system against ROS, these antioxidant defenses are not fully effective during sun exposure and weaken over time. Photoaging of the skin is characterized by the development of pigmentary disorders, such as actinic lentigos (AL), as well as benign skin tumors such as actinic keratosis (AK), both of which are target pathologies for this study.

AL usually occur in the elderly. They are usually benign but can cause aesthetic problems. They are commonly seen on the hands but can appear on all areas of the body, especially on sun-exposed areas such as the face, back, arms, feet, shoulders and skull. There are different treatment approaches, including physical therapy such as laser therapy, pulsed light, chemical peeling, bleaching and cryotherapy or topical therapy such as hydroquinone (HQ). Although topical therapies are generally more time consuming compared to physical therapies, patients can control their own treatment and side effects can be decreased.

AK is a very common skin lesion caused by chronic sun damage that typically measure less than 1 cm in diameter. KA is considered a premalignant epithelial skin lesion that may progress to squamous cell carcinoma. For this reason, all KA should be treated and clinical follow-up is recommended. The goals of treatment are: (i) to clinically eradicate obvious and subclinical lesions, (ii) to prevent their progression to EC, and (iii) to reduce the number of relapses and consequently increase the quality of life of patients.

Medical treatment with antioxidant properties/actions that would allow the reduction of damaged cells seems to play a role in both the prevention and treatment of AL and KA (Nashan et al., 2013).

In addition, a paper published in early 2020 highlighted a major role for carbonylation in the progression of this type of skin lesion (Tramutola et al., 2020). Based on these elements, we hypothesize that our cosmetic active ingredient - MRB - which has antioxidant activity and a specific and original chaperone effect giving it a strong capacity to fight against protein carbonylation- will be effective in the treatment of photo-induced signs of aging: keratoses and actinic lentigo, by a mechanism that acts on the oxidative stress pathway and the maintenance of cellular proteostasis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 5 actinic lentigos and 3 actinic keratoses of grade 1 or 2 on each hemi-face of the face and/or hemi-cranium (in men with baldness)
* Phototype I to III
* Patients with free, informed, written consent to participate in the study.
* Women unable to conceive or women of childbearing potential with a negative urine pregnancy test and using contraception

Exclusion Criteria:

* Subjects with less than 5 actinic lentigos or less than 3 actinic keratoses of grade 1 or 2 on each hemiface of the face and/or skull (for men with baldness)
* Phototype IV to VI
* Immunocompromised subject
* Subjects with a history of skin carcinoma in the treated areas
* Subjects using another active treatment for actinic keratoses or lentigos (or having used one in the past 3 months)
* Subjects unable to understand the information (due to language or psychiatric reasons)
* Subjects without social insurance
* Pregnant women
* Breastfeeding women
* Women of childbearing age without contraception
* Subjects under legal protection measures
* Subjects unable to express their consent
* Subjects under legal protection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate MRB 0.3% serum effectiveness after 6 months of treatment on 2 early clinical markers of photoinduced cutaneous aging: actinic lentigo and actinic keratosis | 6 months
  The primary endpoint will be the decrease at 6 months from baseline in the overall score determined by the sum of the total number of actinic lentigos and actinic keratoses on each hemi-face, one receiving MRB 0.3% serum and the other a placebo serum. For men with baldness, the evaluation could be performed on each hemi-skull and/or each hemi-face.
  The counting of the two types of lesions will be done by simple dermatological examination.

SECONDARY OUTCOMES:
To evaluate 0.3% MRB serum effectiveness versus a placebo serum at inclusion, 1, 3 and 6 months of treatment on the evolution of actinic lentigos on each hemi- face and/or skull | 1, 3 and 6 months
  Assessment at inclusion (T0), after 1 month, 3 months and 6 months of treatment of the number of actinic lentigos on each hemiface and/or hemiskull (in men with baldness) treated with MRB serum 0.3% and placebo serum respectively. The counting of the lesions will be done by simple dermatological examination.
To evaluate 0.3% MRB serum effectiveness versus a placebo serum at inclusion, 1, 3 and 6 months of treatment on the evolution actinic keratoses on each hemi-face/skull | 1, 3 and 6 months
  Assessment at inclusion (T0), after 1 month, 3 months and 6 months of treatment of the number of actinic keratoses on each hemi-facial and/or hemi-cranial area (in men with baldness) treated with MRB 0.3% serum and placebo serum respectively. The counting of the lesions will be done by simple dermatological examination.
To evaluate 0.3% MRB serum effectiveness versus a placebo serum at inclusion, 1, 3 and 6 months of treatment on the grade of actinic keratoses on each hemi-face/skull | 1, 3 and 6 months
  Assessment at inclusion (T0), after 1 month, 3 months and 6 months of treatment of the grade of actinic keratosis defined by the AK-FAS (Actinic Keratosis Field Assessment Scale)
To evaluate in the long term, at 9 and 12 months, on the whole face and/or skull the effect of a MRB 0.3% serum on actinic lentigos and actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on the whole face and/or skull of the overall score determined by the sum of the total number of actinic lentigos and actinic keratoses on the whole face and/or skull. The counting of the two types of lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on the whole face and/or skull the effect of a MRB 0.3% serum on actinic lentigos | 9 and 12 months
  Assessment after 9 months and 12 months on the whole face and/or skull of the number of actinic lentigos.
  The counting of the lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on the whole face and/or skull the effect of a MRB 0.3% serum on actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on the whole face and/or skull of the number of actinic keratoses.
  The counting of the lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on the whole face and/or skull the effect of a MRB 0.3% serum on the grade of actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on the whole face and/or skull of the AK-FAS grade of actinic keratosis.
To evaluate in the long term, at 9 and 12 months, on each hemi-face and/or skull the effect of a MRB 0.3% serum on actinic lentigos | 9 and 12 months
  Assessment after 9 months and 12 months on each hemi-face and/or hemi-skull (in men with baldness) of the number of actinic lentigos.
  The counting of the lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on each hemi-face and/or skull the effect of a MRB 0.3% serum on actinic lentigos and actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on each hemi-face and/or hemi-skull (in men with baldness) of the overall score determined by the sum of the total number of actinic lentigos and actinic keratoses on each hemi-face.
  The counting of the two types of lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on each hemi-face and/or skull the effect of a MRB 0.3% serum on actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on each hemi-face and/or hemi-skull (in men with baldness) of the number of actinic keratoses.
  The counting of the two types of lesions will be done by simple dermatological examination.
To evaluate in the long term, at 9 and 12 months, on each hemi-face and/or skull (in men with baldness) the effect of a MRB 0.3% serum on the grade of actinic keratoses | 9 and 12 months
  Assessment after 9 months and 12 months on each hemi-face and/or hemi-skull (in men with baldness) of the AK-FAS grade of actinic keratosis.
To evaluate at each visit, the tolerance of MRB 0.3% serum versus a placebo serum | 1, 3, 6, 9 and 12 months
  Tolerance assessed at each visit.
  It will be assessed by the investigator during the visits using a 5-point scale (0 = Absent, 1 = Mild, 2 = Moderate, 3 = Severe, 4 = Extreme) evaluating the following parameters:
  1. Erythema
  2. Desquamation
  3. Burning
  4. Pruritus
  5. Stretch A global score of tolerance will be calculated by the sum of the 5 parameters. The global score can vary between 0 and 20.
To evaluate at 6 and 12 months from inclusion, the evolution of a lesioned area and an area of normal skin by confocal microscopy on each hemi-face/skull of 10 volunteer subjects. | 6 and 12 months
  Confocal microscopy of a lesioned area and an area of normal skin: a study of the cells of the epidermis (keratinocytes), the dermis (fibroblasts) and the cellular infiltrate will be performed on a predefined area of each hemi-face/skull of 3 x3 cm at T0 (Inclusion) by Confocal Microscopy with a High Resolution Ultrasound (LC-OCT) and will be repeated at 6 and 12 months in 10 subjects The area will include at least one KA lesion, one lentigo lesion, and the peri-lesional healthy skin area.
To evaluate the satisfaction of the subjects at 6 months (in hemi-face and/or skull), at 9 and 12 months (for the whole face and/or skull and in hemi-face and/or skull) regarding the use of a MRB 0.3 % serum | 6, 9 and 12 months
  Subject satisfaction will be evaluated at 6 months on each hemi-face and/or hemi-skull and at 9 and 12 months on the whole face and/or skull and in hemi-face and/or skull via a satisfaction questionnaire (abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9).
To evaluate the satisfaction of the subjects regardind galenic at 6 months (in hemi-face and/or skull), at 9 and 12 months (for the whole face and/or skull and in hemi-face and/or skull) regarding the use of the applied serums | 6, 9 and 12 months
  Subject satisfaction will be evaluated at 6 months on each hemi-face and/or hemi-skull and at 9 and 12 months on the whole face and/or skull and in hemi-face and/or skull via a questionnaire on the galenic quality of the applied products (texture, ease of application, etc.).
To evaluate the satisfaction of the investigator at 6, 9 and 12 months regarding the products used | 6, 9 and 12 months
  The investigator's satisfaction with the products will be evaluated at 6 months on each hemi-face and/or hemi-skull and at 9 and 12 months on the whole face and/or skull on a 5-point scale:
  1. = Very good effectiveness
  2. = Good effectiveness
  3. = Average effectiveness
  4. = Poor effectiveness
  5. = Not effective at all
To evaluate subjects' compliance with serums application | 1, 3, 6, 9 and 12 months
  Product compliance will be assessed during the visits by weighing the tubes of product collected.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nashan D, Meiss F, Muller M. Therapeutic strategies for actinic keratoses--a systematic review. Eur J Dermatol. 2013 Jan-Feb;23(1):14-32. doi: 10.1684/ejd.2013.1923. PMID 23477760
- [Background] Tramutola A, Falcucci S, Brocco U, Triani F, Lanzillotta C, Donati M, Panetta C, Luzi F, Iavarone F, Vincenzoni F, Castagnola M, Perluigi M, Di Domenico F, Marco F. Protein Oxidative Damage in UV-Related Skin Cancer and Dysplastic Lesions Contributes to Neoplastic Promotion and Progression. Cancers (Basel). 2020 Jan 1;12(1):110. doi: 10.3390/cancers12010110. PMID 31906275